CLINICAL TRIAL: NCT01892930
Title: Immunologic Impact of Stereotactic Body Radiation Therapy (SBRT) in Renal Cell Carcinoma
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Metastatic Kidney Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 212712; NCI-2013-01201 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-06-20; First posted 2013-07-08 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (SBRT, nephrectomy) (Experimental): Patients undergo SBRT on day 1 and undergo partial or radical nephrectomy on day 29.
  Interventions: Radiation: stereotactic body radiation therapy; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Procedure: therapeutic conventional surgery — Undergo partial or radical nephrectomy
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies stereotactic body radiation therapy in treating patients with metastatic kidney cancer undergoing surgery. Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the impact of stereotactic body radiation therapy (SBRT) on the immune system in patients with metastatic renal cell carcinoma (RCC).

SECONDARY OBJECTIVES:

I. Assess changes in immune parameters prior to radiation, post radiation and post nephrectomy.

TERTIARY OBJECTIVES:

I. Assess surgical parameters for partial or radical nephrectomy post SBRT.

OUTLINE:

Patients undergo SBRT on day 1 and undergo partial or radical nephrectomy on day 29.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Have metastatic RCC with primary tumor in place
* Must be surgical candidates as deemed fit by surgeon
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Patients of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Radiation to primary tumor prior to enrollment in this study
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive treatment
* Received an investigational agent within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting a partial nephrectomy in patients with no prior stereotactic radiation for kidney cancer | Up to 30 days post-treatment

SECONDARY OUTCOMES:
Toxicity analysis assessed by the CTEP Version 4 of the NCI Common Terminology Criteria for Adverse Events (CTCAE) | Up to 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schwaab, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Singh AK, Winslow TB, Kermany MH, Goritz V, Heit L, Miller A, Hoffend NC, Stein LC, Kumaraswamy LK, Warren GW, Bshara W, Odunsi K, Matsuzaki J, Abrams SI, Schwaab T, Muhitch JB. A Pilot Study of Stereotactic Body Radiation Therapy Combined with Cytoreductive Nephrectomy for Metastatic Renal Cell Carcinoma. Clin Cancer Res. 2017 Sep 1;23(17):5055-5065. doi: 10.1158/1078-0432.CCR-16-2946. Epub 2017 Jun 19. PMID 28630212